CLINICAL TRIAL: NCT02495649
Title: Evaluation of Myocardial Sympathetic Denervation in Parkinson's Disease Using [18F]FDOPA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, Michal Roll PhD,MBA, DIRECTOR R&D devition, Tel-Aviv Sourasky Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TASMO-15-ES-0606-14-TLV-CTIL
Record Dates: First submitted 2015-06-03; First posted 2015-07-13 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Parkinson
MeSH Terms: interventions — fluorodopa F 18; Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [18F]-DOPA (Other): evaluate the added value of PET-CT with [18F]-DOPA tracer for Assessment of the Myocardial Sympathetic Denervation in patients with or suspected with Parkinson's disease.
  Interventions: Other: [18F]-DOPA; Device: PET-CT

INTERVENTIONS:
Other: [18F]-DOPA — To evaluate the feasibility of PET-CT with [18F]-DOPA to assess the myocardial sympathetic denervation in patients with or suspected with Parkinson's disease
Device: PET-CT — To evaluate the feasibility of PET-CT with [18F]-DOPA to assess the myocardial sympathetic denervation in patients with or suspected with Parkinson's disease

SUMMARY:
The purpose of this study is to evaluate the added value of PET-CT with [18F]FDOPA tracer for Assessment of the Myocardial Sympathetic Denervation in patients with or suspected with Parkinson's disease.

The investigators expect to see normal values of uptake ratio of [18F]FDOPA , in patients with no synuclein underline pathology or previously known cardiovascular disease (no history of high blood pressure or take medications that influence the sympathetic system- exclusion criteria). Low values of uptake ratio is presumed to be found in patients diagnosed with Parkinson's disease or other synuclein pathology.

The expected normal ratio of Heart/liver uptake values will be determined from scans of patients refered to [18F]FDOPA scan and were found to have normal [18F]FDOPA scan of the basal ganglia and no cardiovascular diseases.

DETAILED DESCRIPTION:
L-3,4-dihydroxy-6-[18F]fluoro-phenylalanine ([18F]FDOPA) might be a useful tracer for assessing myocardial sympathetic denervation in Parkinson's disease (PD) Patients. Compared to the routinely used I123 MIBG scan, [18F]FDOPA seems to have an advantage for the following reasons:

1. meta-iodobenzylguanidine (MIBG) is a false analog of norepinephrine while [18F]FDOPA is the radiolabelled form of DOPA, a direct precursor of dopamine which is subsequently converted to norepinephrine
2. 123I MIBG, un-like norepinephrine, dose not undergo intracellular metabolism (19) while [18F]FDOPA undergo complex intracellular metabolism (17)
3. Studies have shown that I123 MIBG reuptake is almost exclusive by uptake mechanism 1. Uptake-2 mechanism of 123I-MIBG by the myocardium is not significant. Reuptake of norepinephrine (NE) in the synaptic cleft and is mainly by uptake 1 system but also in small amount by uptake 2 systems. The investigators assumption is that this double mechanism of reuptake will increase the concentration of [18F]FDOPA for better imaging

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Signed Informed Consent
3. Patients referred for F-dopa scan of basal ganglia in the evaluation of Parkinson's disease or other extra pyramidal motor disorders.
4. Patients diagnosed with Parkinson's disease.

Exclusion Criteria:

1. Age < 18
2. Previous diagnosed Heart Disease.
3. History of High blood pressure.
4. On medications that influence the sympathetic system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-08 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
The uptake of [18F]FDOPA will be measured by the ratio between the uptake in the heart and the uptake in the liver. | paitents will be scanned in PET- CT scaner for 10 minutes
  The uptake value of [18F]FDOPA will be measured by the ratio of standard uptake value (SUV) in the heart and the SUV in the liver.
  Normal uptake will be calculated by the mean uptake ratio in the healthy population (plus minus standard deviation) and used to compare to patients with abnormal [18F]FDOPA scan of the basal ganglia.

CONTACTS AND LOCATIONS:
Overall Officials: Einat Even Sapir, Phd, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Sourasky Medical Center, Tel Aviv, Israel